CLINICAL TRIAL: NCT03634020
Title: Evaluation of a Thin Strut Metallic Coronary Device: the Elixir DynamXTM Sirolimus Eluting Coronary Bioadaptor System
Brief Title: DynamX Sirolimus Study Sirolimus Eluting Coronary Bioadaptor System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1801
Record Dates: First submitted 2018-08-01; First posted 2018-08-16 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: prospective, consecutive enrollment, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DynamX Sirolimus-eluting Coronary Bioadaptor System (Experimental): 2.5 - 3.5mm 14mm, 18mm and 28mm
  Interventions: Device: DynamX Sirolimus-eluting Coronary Bioadaptor System

INTERVENTIONS:
Device: DynamX Sirolimus-eluting Coronary Bioadaptor System — de novo native coronary artery lesions

SUMMARY:
To confirm the safety and performance of the DynamX Sirolimus-eluting Coronary Bioadaptor System (SECBS) in de novo native coronary artery lesions using clinical and imaging endpoints. Clinical follow-up will be conducted in all patients at 30 days, 6 and 12 months. Imaging follow-up will be conducted at 6 months.

DETAILED DESCRIPTION:
The DynamX Sirolimus Study is a prospective, consecutive enrollment, single-arm study designed to enroll up to 30 patients requiring treatment of up to two de novo lesions ≤ 24 mm in length in vessels ≥ 2.5 mm and ≤ 3.5 mm in diameter.

One or two designated target lesions, located in separate epicardial vessels (RCA, LCX or LAD), and meeting the inclusion/exclusion criteria may be treated with the DynamX SECBS. Alternatively, one target lesion may be treated with the DynamX SECBS after successful, uncomplicated treatment of a non-target lesion, located in a separate epicardial vessel, with any commercially-available DES. Acceptable example: non-target RCA lesion and LAD target lesion. Not acceptable example: LAD non-target lesion and 1st diagonal target lesion.

The primary safety endpoint is Target Lesion Failure at 6 months. TLF is a composite endpoint defined as cardiac death, target vessel MI, and clinically-indicated target lesion revascularization The primary efficacy endpoint is late lumen loss at 6 months, assessed by angiography Additional secondary safety and effectiveness endpoints will be evaluated at 30 days, 6 and 12 months Using visual assessment, the target lesion must measure ≥ 2.5 mm and ≤ 3.5 mm in diameter and ≤ 24 mm in length able to be covered by a single DynamX Sirolimus Bioadaptor including 2 mm of healthy vessel on either side of the planned treatment area.

The patient will be eligible for stent (also called bioadaptor) implantation only after satisfactory lesion pre-dilatation defined as: ≥ TIMI 2 flow, and no dissection greater than Grade B (NHLBI) able to be covered with a single DynamX SECBS

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age
2. Patient is able to understand the risks, benefits and treatment alternatives of receiving the DynamX Sirolimus Eluting CBS and provide written informed consent, as approved by the NZ Ethics Committee, prior to any clinical study-related procedure
3. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
5. Women of childbearing potential with a negative pregnancy test within 7 days and women who are not pregnant or nursing
6. Patient must agree to undergo all clinical study required follow up visits, angiograms, and imaging testing
7. Patient must agree not to participate in any other clinical research study for a period of one year following the index procedure Angiographic inclusion criteria- Target Lesion/Vessel
8. Target lesion(s) must be located in a native coronary artery with a vessel diameter of ≥ 2.5 and ≤3.5 mm assessed visually or by online QCA
9. Target lesion(s) must measure ≤ 24 mm in length
10. Target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 90% with a TIMI flow of ≥ 2. When two target lesions are treated, they must be located in separate major epicardial vessels
11. The lesion(s) must be successfully pre-dilated (less than 35% DS) prior to enrollment
12. The target lesion length is 24 mm and able to be covered by a single DynamX Sirolimus Bioadaptor with 2 mm of healthy vessel on either side of planned implantation site
13. Treatment of a single, non-target lesion located in a separate major epicardial vessel

Exclusion Criteria:

1. Patient has a diagnosis of ST elevation myocardial infarction (STEMI) within 72 hours preceding the index procedure, and CK and CK-MB have not returned within normal limits at the time of procedure
2. Patient requires the use of rotational atherectomy during the index procedure
3. Patient has current unstable ventricular arrhythmias
4. Patient has a known left ventricular ejection fraction (LVEF) < 30%
5. Patient has received a heart transplant or any other organ transplant or is on a waiting list for an organ transplant
6. Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
7. Patient is receiving immunosuppression therapy, other than steroids or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
8. Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, prasugrel or ticagrelor, Sirolimus, CoCr alloys, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
9. Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel or other P2Y12 inhibitors.
10. Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented liver disease.
11. Patient has severe renal dysfunction (CKD IV or V, eGFR <30) or is on dialysis.
12. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
13. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
14. Patient has had a significant GI or urinary bleed within the past six months
15. Patient has a condition that precludes safe 6 French sheath insertion; or other medical conditions or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or associated with a limited life expectancy (i.e., less than one year)
16. Patient is already participating in another clinical study which has not reached the primary endpoint (long-term follow-up is not an exclusion) Angiographic Exclusion Criteria Target Lesion/Vessel

1. Target/Vessel / Target lesion(s) meets any of the following criteria:

1. Aorto-ostial location
2. Left main location
3. Located within 5 mm of the origin of the LAD or LCX
4. Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
5. Lesion involving a bifurcation with a side branch >2mm in diameter
6. Previous placement of a stent within 10 mm of the target lesion
7. Total or sub-total occlusion (TIMI flow ≤1)
8. The proximal target vessel or target lesion is severely calcified by visual assessment, or the lesion prevents full pre-dilatation balloon expansion
9. Previous intervention restenosis 2. The target vessel contains visible thrombus 3. Another clinically-significant lesion (>50%) is located in the same major epicardial vessel as the target lesion 5. Target vessel was previously treated with any type of PCI < 6 months prior to index procedure 6. Non-Target vessel was previously treated with any type of PCI < 30 days prior to the index procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Target Lesion (s) Failure | 6 months
  composite endpoint of cardiac death, target vessel MI and clinically-indicated TLR

SECONDARY OUTCOMES:
Target Lesion (s) Failure | 1 month
  composite endpoint of cardiac death, target vessel MI and clinically-indicated TLR
Target Lesion (s) Failure | 12 month
  composite endpoint of cardiac death, target vessel MI and clinically-indicated TLR
cardiac death | 1 month
  death from a cardiac cause
Cardiac Death | 6 months
  death from a cardiac cause
Cardiac Death | 12 months
  death from a cardiac cause
Non-Cardiac Death | 1 month
  death from a non-cardiac cause
Non-Cardiac Death | 6 months
  death from a non-cardiac cause
Non-Cardiac Death | 12 months
  death from a non-cardiac cause
myocardial infarction | 1 month
  all
myocardial infarction | 6 months
  all
myocardial infarction | 12 months
  all
myocardial infarction | 1 month
  related to the target vessel
myocardial infarction | 6 months
  related to the target vessel
Target Lesion Revascularization | 1 month
  Clinically indicated repeat intervention within the target lesion
Target Lesion Revascularization | 6 months
  Clinically indicated repeat intervention within the target lesion
Target Lesion Revascularization | 12 months
  Clinically indicated repeat intervention within the target lesion
Target Vessel Revascularization | 1 month
  Clinically indicated repeat intervention within the target vessel
Target Vessel Revascularization | 6 months
  Clinically indicated repeat intervention within the target vessel
Target Vessel Revascularization | 12 months
  Clinically indicated repeat intervention within the target vessel
Device Thrombosis | 1 month
  definite and probable as classified by an Academic Research Consortium
Device Thrombosis | 6 months
  definite and probable as classified by an Academic Research Consortium
Device Thrombosis | 12 months
  definite and probable as classified by an Academic Research Consortium

OTHER OUTCOMES:
Qualitative coronary angiography | 6 months
  in-device late lumen loss
Intravascular ultrasound imaging | 6 months
  Change in mean lumen area from post-procedure to 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (7):
- New Zealand (7):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No